CLINICAL TRIAL: NCT01889056
Title: Non-erythroid Effects of Erythropoietin on Cognitive Function and Exercise Capacity in Humans
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EPOPERF CH12
Record Dates: First submitted 2013-02-26; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Erythropoietin; Cognition; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Erythropoietin; epoetin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Erythropoietin (Epoetin beta) (Experimental): Short infusion of 60.000 IU Epoetin beta in 0.9% sodium chloride solution (250 ml)
  Interventions: Drug: Erythropoietin (Epoetin beta)
- 0.9% sodium chloride solution (Placebo Comparator): Short infusion of 0.9% sodium chloride solution (250 ml)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythropoietin (Epoetin beta)
  Other Names: Recormon
  Arms: Erythropoietin (Epoetin beta)
Drug: Placebo — 0.9% sodium chloride solution
  Arms: 0.9% sodium chloride solution

SUMMARY:
The blood hormone Erythropoietin (Epo) is not only produced by the kidneys but also by the brain, especially under hypoxic conditions. It has been shown in animal studies and human studies that Epo has neuroprotective properties. Furthermore, there is scientific evidence for central modulatory effects of Epo in the brain but high dose of Epo is needed to overcome the blood brain barrier. In a double blind placebo controlled crossover study we will investigate the effects of a single high dose of Epo on cognitive function and exercise capacity in healthy subjects. The subjects will receive a single high dose of Epo (60.000 IU) and will perform a computerized cognitive test battery, a breathing test, a maximal exercise capacity test (VO2max), and a time trial (TT) 24 hours after the treatment. The primary outcome of the study will be the cognitive function.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Healthy Subjects;
* Age between 18 to 35 years;
* Normal body weight (body mass index of >= 18.5 kg/m2 <= 24.9 kg/m2);
* Nonsmokers (>= 1 year);
* VO2max of <= 55 ml/kg/min for females and <= 60 ml/kg/min for males;

Exclusion criteria:

* Persons with abnormal Serum Ferritin levels according to gender dependent reference values of GCP-certificated laboratory;
* Persons with pre-existing genetic hemostatic disorders (Factor V Leiden mutation, Prothrombin mutation);
* Persons which are at risk of deep venous thrombosis (e.g. history of venous thromboembolic events);
* Persons with a hematocrit value of > 55%;
* Persons being exposed to prolonged (>= 5 days) high altitude (>= 2500m above Normal Null) <= 6 months prior the beginning of the study;
* Persons not willing to maintain their living conditions during the study period (e.g. preparing for a certain competition);
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product;
* Pregnant or breast feeding women;
* Intention to become pregnant during the course of the study;
* Lack of safe contraception;
* Treatment with other investigational products;
* Known or suspected non-compliance, drug or alcohol abuse;
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders;
* Participation in another study with investigational drug within the 30 days preceding and during the present study;
* Enrolment of the investigator, his/her family members, employees and other dependent persons;

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | 1 year
  The following parameters of cognitive function will be tested via computer-based cognitive testing (Units: Scores, Percent Correct, Response time):
  * Working memory capacity
  * Executive function
  * Processing speed

SECONDARY OUTCOMES:
Exercise Capacity | 1 year
  Evaluation of exercise capacity via specific exercise tests:
  * VO2max test
  * 20-minutes time trial (TT)

OTHER OUTCOMES:
Subjective Well-Being | 1 year
  Evaluation of subjective well-being via:
  * Questionnaires
  * Visual Analog Scales

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, Prof MD, Principal Investigator — University Hospital Zurich, Medical intensive care unit
Locations (1):
- University Hospital Zurich, Medical intensive care unit, Zurich, Canton of Zurich, Switzerland